CLINICAL TRIAL: NCT04166032
Title: Validation Study for the Alertgy Non-invasive Continuous Glucose Monitor
Brief Title: Validation Study for the Alertgy Non-invasive Continuous Glucose Monitor (ANICGM)
Status: Completed | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Alertgy (Industry)
Responsible Party: Principal Investigator, M. Cecilia Lansang, MD, Professor of Medicine, Endocrinology Staff Physician, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 18-1385
Record Dates: First submitted 2019-11-13; First posted 2019-11-18 (Actual); Results first posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-10

CONDITIONS: Type 2 Diabetes
Keywords: glucose monitor
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- ANICGM (Experimental): non-invasive continuous glucose monitoring device
  Interventions: Device: Alertgy non-invasive continuous glucose monitoring device (ANICGM)

INTERVENTIONS:
Device: Alertgy non-invasive continuous glucose monitoring device (ANICGM) — Alertgy non-invasive continuous glucose monitoring device (ANICGM)

SUMMARY:
Diabetes mellitus (DM) affects 30 million people in the United States. To achieve glucose control, most patients are prescribed glucose meters by their physicians. Obtaining glucose levels in this manner necessitates cleaning the fingers, attaching a lancet to a device (or simply using a lancet if a device is not available), pricking the finger with a lancet, placing a drop blood on a strip, and awaiting the readout that results after some chemical reactions. Thereafter, the lancet has to be disposed of in a safe receptacle and the finger has to be blotted to stop the blood from oozing.

The anxiety, pain, and tedious process have led researchers to develop other means of checking glucose levels. There are now continuous glucose monitoring systems (CGMS) that entail inserting a subcutaneous sensor that sends readings through a transmitter. These CGMs may or may not need calibration with a fingerstick glucose reading, and the subcutaneous sensor still has to be changed every 10 -14 days.

The Alertgy non-invasive continuous glucose monitor (ANICGM) is a device that does not entail any subcutaneous insertion of a sensor. It is strapped on to the wrist, and glucose readings are given based on subcutaneous signals. In 2001, a non-invasive device called Glucowatch Biographer was introduced that also involved subcutaneous signals without needing a subcutaneous insertion. However, for various reasons such as long calibration period and reading inaccuracies, the product did not take off. The ANICGM is a promising device that might overcome the limitations of existing and previous methods of non-invasive glucose measurement.

DETAILED DESCRIPTION:
The ANICGM uses a weak electromagnetic field generated by its wrist band sensor to look into the body to produce a spectrum that provides a measurement of blood glucose present in the wrist area of the body. The core sensing technology used is dielectric spectroscopy, and has been shown capable of measuring blood glucose, non-invasively, in a laboratory environment. The system uses proprietary and patented dielectric materials and signal processing to enhance performance in both selectivity and sensitivity for blood glucose measurement.

Much like how a MRI uses a strong magnetic field and its interaction with the body to create a picture of what is inside, the ANICGM uses a safe weak low frequency radiofrequency field to take a picture of a person's chemical spectrum, some of it specific only to blood glucose.

The device sends and receives back signals from the wrist area that are used to generate a dielectric spectrum once every 6 seconds. The POC BG using the Accuchek Inform II will be used to provide calibration values for the ANICGM every 5 minutes in mg/dL, during the calibration process. The POC BG levels will be entered into the Alertgy laptop and a proprietary calibration program will be used to analyze the spectral data collected and will generate a calibration algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes on diet or on pharmacologic treatment for diabetes
* Hemoglobin A1c between 7.5 - 10.0%
* Age 18 - 75 years old

Exclusion Criteria:

* Patients taking prandial insulin
* Fasting blood glucose by fingerstick of < 70 mg/dL or >250 mg/dL
* Pregnancy
* End stage renal disease
* Decompensated or acute heart failure
* Medications that may cause false readings with glucose meters: acetaminophen, ascorbic acid, dopamine, maltodextrin, mannitol
* Conditions that limit the ANICGM such as lesions on the forearms
* Other conditions that the investigator deems will affect the conduct of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-05-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ANICGM
Started | 15
Completed | 14
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | ANICGM
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Mean Absolute Relative Difference (MARD) of Glucose Values Between the ANICGM and FDA-approved Glucose Monitoring Device
Description: Hypothesis is that ANICGM device will perform similarly as other blood glucose monitoring devices Mean absolute relative difference (MARD) is computed by taking the arithmetic mean of the absolute relative differences between the ANICGM system measures and the reference standard FS BG, which serves as the denominator of the calculation. The MARD is expressed as a percentage, and a lower MARD signifies better concordance between the two measurements.
Time Frame: 2 time points taken over 2 separate days respectively, over a span of up to 14 days
Measure: Mean (95% Confidence Interval); unit: percentage difference
Arm/Group | ANICGM
Number analyzed (Participants) | 15
percentage difference
  Day 2 | 18 [12.8 to 42.2]
  Day 3 | 15 [12.3 to 18.4]
Statistical Analysis 1: Comparison: ANICGM; Test type: Other; p = 0.210, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 3 months
Description: No adverse events reported
Arm/Group | ANICGM
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Company will review any publication submission within 30 days of estimated due date. If CCF does not hear from company we are to assume we are free to publish. If company identities patentable information they can request for CCF to withhold submission for 90 days.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/32/NCT04166032/Prot_SAP_000.pdf